CLINICAL TRIAL: NCT01397864
Title: C1 Inhibitor Treatment Registry to Assess the Safety and Immunological Profile of Ruconest in the Treatment of HAE Attacks
Brief Title: C1 Inhibitor Registry in the Treatment of Hereditary Angioedema (HAE) Attacks
Status: Completed | Type: Observational
Sponsor: Pharming Technologies B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: C1 1412
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary Angioedema; HAE; Angioedema; Recombinant C1 Inhibitor; rhC1INH; registry
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema | interventions — conestat alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hereditary Angioedema
  Interventions: Drug: rhC1INH or pdC1INH

INTERVENTIONS:
Drug: rhC1INH or pdC1INH — C1 inhibitor, either plasma-derived (pdC1INH) or the recombinant human form (Ruconest)
  Other Names: Ruconest

SUMMARY:
This is a non-interventional treatment Registry of Hereditary Angioedema (HAE) patients treated with C1 inhibitor, either plasma-derived (pdC1INH) or the recombinant human form (rhC1INH / Ruconest), to observe adverse events and insufficient efficacy, and to assess the immunological profile following single and repeated treatment with Ruconest.

DETAILED DESCRIPTION:
see below

ELIGIBILITY:
Inclusion Criteria:

* Decision to treat the HAE patient with C1 inhibitor (either Ruconest or pdC1INH)
* Patients must give written informed consent

Exclusion Criteria:

* A diagnosis of acquired C1INH deficiency (AAE)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The aim is to recruit 300 patients treated with Ruconest. Additionally, the study will continue until 100 patients have been exposed to Ruconest for at least 3 attacks. Enrolment in the pdC1INH arm will be unrestricted.
Sampling Method: Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
The primary objective is to observe the adverse event profile and insufficient efficacy, following single and repeated treatment with Ruconest or pdC1INH of acute angioedema attacks | December 2019

SECONDARY OUTCOMES:
To assess the immunological profile of Ruconest (for suspected hypersensitivity or suspected neutralizing antibodies) | December 2019

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Relan, MD, Study Director — Pharming Technologies BV
Locations (17):
- UMHAT Alexandrovska EAD, Sofia, Bulgaria
- Croatia (3):
  - KBC Split, Split
  - General Hospital Sibenik, Šibenik
  - CHC Sestre milosrdnice, Zagreb
- Faculty Hospital by St. Anna Brno, Brno, Czechia
- Hospital A Michallon, CHU Grenoble, La Tronche, France
- Charite Universitatsmedizin Berlin, Berlin, Germany
- Semmelweis University, 3rd Department of Internal Medicine, Budapest, Hungary
- Ospedale Luigi Sacco, Milan, Italy
- PHI University Clinic of Dermatology, Skopje, North Macedonia
- Norway (2):
  - Alesund Hospital, Ålesund
  - Stavanger University Hospital, Stavanger
- University Hospital Krakow, Krakow, Poland
- Slovakia (2):
  - Bratislava University Hospital, Bratislava
  - University Hospital Martin, Martin
- University Clinic Golnik, Golnik, Slovenia
- Ryhof County Hospital, Jönköping, Sweden